CLINICAL TRIAL: NCT00002973
Title: Phase II Evaluation of IV Melphalan (L-PAM) and Whole Body Hyperthermia (WBH) for Malignant Melanoma
Brief Title: Melphalan and Whole-Body Hyperthermia in Treating Patients With Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000065487; WCCC-CO-9571; NCI-G97-1216
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Melphalan; Diathermy

INTERVENTIONS:
Drug: melphalan
Procedure: hyperthermia treatment

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Hyperthermia therapy kills tumor cells by heating them to several degrees above body temperature. Combining hyperthermia with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of melphalan and whole-body hyperthermia in treating patients with advanced melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the combination of 41.8 degrees Celsius whole body hyperthermia (WBH) and melphalan (L-PAM) in patients with advanced melanoma. II. Assess the efficacy of this combination of therapy. III. Assess the clinical toxicity of WBH and L-PAM in these patients. IV. Obtain pilot data on the effect of WBH and L-PAM on cytokine induction in these patients.

OUTLINE: The combination of whole body hyperthermia (WBH) and melphalan (L-PAM) is administered on week 1. The infusion of L-PAM is administered at a constant rate over approximately 10 minutes, beginning 20 minutes after achieving target temperature of 41.8 degrees Celsius by esophageal or axillary temperature probe. WBH is continued for an additional 40 minutes for a total of 60 minutes. On week 5 or 6, patients receive another combination of WBH and L-PAM. Disease status is reevaluated at least every 2 courses. Patients without progressive disease continue therapy of WBH and L-PAM every 4 weeks for a maximum of 6 courses.

PROJECTED ACCRUAL: Approximately 34 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced melanoma beyond hope of surgical cure or metastatic disease Tumors must be refractory to all known forms of effective therapy No CNS tumor involvement No major liver involvement (more than 33% replacement of liver by tumor)

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: WBC greater than 3,000/mm3 Absolute granulocyte count at least 1,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Alkaline phosphatase no greater than 3 times normal SGOT no greater than 3 times normal Protein no less than 15% below lower limit of normal Renal: BUN less than 30 mg/dL Creatinine less than 1.5 mg/dL OR Creatinine clearance no less than 60 mL/min Calcium no greater than 11.0 mg/dL Sodium 130-150 mEq/L Potassium 3.0-5.0 mg/dL Cardiovascular: No organic heart disease, including: - coronary artery disease - history of angina - history of dysrhythmia requiring ongoing medical intervention - uncontrolled hypertension - patients requiring beta blockers Neurologic: No moderate or severe peripheral neuropathy No history of severe emotional instability by psychiatric history Pulmonary: FEV1 at least 60% of predicted Maximum voluntary volume at least 60% of predicted Partial pressure of oxygen at least 60 OR Oxygen saturation at least 90% Other: No history of secondary primary cancer which conceivably could be active No active nonmalignant gastric and/or duodenal ulcer No serious infection requiring hospitalization within the previous 14 days No history of hepatitis related to general anesthesia No history of allergy to lidocaine or related compounds No development of malignant hyperthermia after general anesthesia No unexplained persistent fever Not pregnant or nursing

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since biologic therapy Chemotherapy: At least 8 weeks since nitrosoureas (e.g., lomustine, carmustine, mitomycin) At least 4 weeks since any other chemotherapy Recovered from all toxic effects No concurrent chemotherapy Endocrine therapy: At least 4 weeks since endocrine therapy No concurrent hormonal therapy Radiotherapy: At least 4 weeks since radiotherapy No prior irradiation of more than 25% of the marrow Surgery: Not specified Other: No concurrent nonsteroidal antiinflammatory agents or aspirin

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 1995-12; Primary Completion 2000-05 (Actual); Study Completion 2000-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. I. Robins, MD, PhD, Study Chair — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin, United States